CLINICAL TRIAL: NCT06208527
Title: The NADage Study: a Randomized Double-blind Trial of NAD Replenishment Therapy on Aging
Brief Title: The NADage Study: Nicotinamide Riboside Replenishment Therapy Against Functional Decline in Aging
Acronym: NADage
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Haukeland University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2023/680827
Record Dates: First submitted 2023-11-14; First posted 2024-01-17 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2024-12

CONDITIONS: Frailty; Frail Elderly Syndrome; Frailty Syndrome; Aging
Keywords: Frailty; Nicotinamide Riboside; NR; Nicotinamide adenine dinucleotide; NAD; Frail; Aging; Functional decline
MeSH Terms: conditions — Frailty | interventions — nicotinamide-beta-riboside

STUDY DESIGN:
Intervention Model Description: Randomized double-blinded placebo-controlled study with a duration of 1 year. 100 participants randomized to either Placebo (n=50) or NR 2000 mg (n=50).
Who Masked: Participant, Care Provider, Investigator
Masking Description: Participants and all care providers and investigators are blinded during the trial and during data analysis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Placebo group (Placebo Comparator): Placebo, no active ingredients. Administered in tablet form twice daily for the duration of the trial (1 year).
  Interventions: Other: Placebo
- NR group (Experimental): Nicotinamide Riboside (NR) administered in doses of 1000 mg twice daily for the duration of the trial (1 year).
  Interventions: Dietary Supplement: Nicotinamide Riboside (NR)

INTERVENTIONS:
Dietary Supplement: Nicotinamide Riboside (NR) — A total of 2000 mg NR is administered daily for 1 year.
  Arms: NR group
Other: Placebo — Placebo tablet identical in taste, shape and appearance to NR tablets.
  Arms: Placebo group

SUMMARY:
This clinical study, designed as a double-blind, randomized, placebo-controlled trial, aims to investigate the potential of nicotinamide riboside (NR) to decelerate functional decline in the elderly frail population. In animal studies, NR, which is converted to nicotinamide adenine dinucleotide (NAD), has shown potential as a neuroprotective agent, with indications of protection against amyotrophic lateral sclerosis (ALS), Alzheimer's dementia, and Parkinson's disease. Furthermore, aging is commonly associated with decreased tissue NAD levels, a phenomenon linked to premature aging and a spectrum of age-related disorders, including cardiovascular diseases and cancers. Existing preclinical and clinical research highlights the promise of NAD replenishment through enhanced DNA repair, sirtuin activity, and improved mitochondrial function. The research center has conducted two phase II clinical trials on NR for Parkinson's disease (NAD-PARK and NR-SAFE), administering up to 3000 mg of NR daily. These trials have shown promising results, indicating NR's potential as a treatment that may alter the course of the disease and possibly as neuroprotective treatment in Parkinson's disease.

The NAD age trial primarily aims to determine:

* The efficacy of NAD therapy in improving clinical symptoms of frailty, evaluated through standardized physical and cognitive function tests.
* The safety of administering 2000 mg NR daily in an elderly frail population.

The study will include 100 individuals, classified as frail based on the Fried Frailty Phenotype. Participants will be randomly assigned to receive either 2000 mg of NR daily or a placebo. Over a 52-week period, participants will undergo:

* Clinical evaluations, including actigraphy and questionnaires.
* Cognitive assessments.
* Bio sampling.
* Magnetic resonance imaging (MRI).
* Positron emission tomography (FDG-PET) scanning.

The outcomes of this study could potentially demonstrate that NR effectively reduces signs of frailty, offering considerable advantages to the individuals affected, their families, and society as a whole.

DETAILED DESCRIPTION:
This study aims to administer 2000 mg of nicotinamide riboside (NR) daily to explore its effects on brain and body metabolism in an elderly, frail population. The research design is a single-center, double-blind, randomized, placebo-controlled approach. Participants will be evenly randomized into two groups in a 1:1 ratio: one to receive a placebo and the other to receive 2000 mg of NR daily. The intervention will last for 52 weeks, during which primary and secondary outcomes will be assessed across and within both groups.

The primary objective is to evaluate the impact of NR on gait speed by comparing the treatment group with the placebo group. Secondary objectives include assessing the safety and tolerability of NR, as well as its clinical effects on physical and cognitive functions, using standardized tests. Furthermore, exploratory objectives will be pursued using various methods such as questionnaires, biosampling, actigraphy, and brain scans. These scans will include 31P-MR-spectrometry to analyze NAD levels in the brain and FDG-PET to assess metabolic network activity. The study will include 100 frail individuals who have provided informed consent. Biological samples to be collected include blood/serum, blood cells, urine, and fecal samples.

Given the previously demonstrated potential of NR in reducing symptoms of Parkinson's disease, this study seeks to expand knowledge of its effects on an elderly, frail population without neurodegenerative disorders. If NR is found to be effective in improving measures of frailty, it could significantly impact societal health and economy, especially considering the extensive socio-economic challenges associated with frailty.

ELIGIBILITY:
Inclusion Criteria:

* Participant must understand the nature of the study and be able to provide written, informed consent.
* Male or female aged ≥ 75 years at baseline.
* Fried Frailty Phenotype score ≥ 3 to identify frail individuals.
* Montreal Cognitive Assessment (MoCA) at screening adjusted to age, gender, and educational level, with a threshold set at the 10th percentile (z-score ≤ -1.28).

Exclusion Criteria:

* Inability to provide informed consent.
* Does not reside in a facility or institution.
* Advanced disability, end-stage disease, presence of severe chronic illness and/or life expectancy of less than a year.
* Inability to complete a 6-minute walk test (6MWT) and/or contraindications to the procedure (history of unstable angina or myocardial infarction within 30 days prior to the test).
* Diagnosis of active malignancy in the last 2 years at baseline (exceptions include non-metastatic skin conditions and non-metastatic and/or treated prostate cancer with stable prostate-specific antigen (PSA) levels in six months prior to baseline). Specific considerations may apply depending on the type of cancer.
* Significant neurological or psychiatric disorders, including but not limited to psychotic disorders, severe bipolar or unipolar depression, multiple sclerosis, uncontrolled seizure conditions, and neurodegenerative disorder.
* A history of cerebrovascular events, excluding transient ischemic attack (TIA) that occurs more than 3 months prior to baseline.
* Hospitalization or major surgery within 3 months prior to baseline.
* Significant changes in medications or treatment plans made less than one month prior to baseline, judged by the site investigator to interfere with the subject's participation in the study.
* Consumption of NAD precursor supplements (e.g., Nicotinamide riboside, nicotinamide mononucleotide or Vitamin B3), or related supplements within 6 months prior to baseline.
* Elective surgeries scheduled during the study duration.
* Concurrent participation in other clinical trials with interventions that could affect frailty measures.
* Any medical history, at the discretion of the investigator, might hinder compliance with study procedures or increase risk to the participant.

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
The between-group (NR vs. Placebo) difference in the change in gait speed. | 52 weeks
  Gait speed is assessed by the 6-minute walk test (6MWT).

SECONDARY OUTCOMES:
Incidence of treatment-emergent adverse events (safety and tolerability). | 52 weeks
  Monitor the frequency and severity of adverse events (AE).
Change in physical performance assessed by the Short Physical Performance Battery (SPPB). | 52 weeks
  SPPB is performed as an objective measurements on balance, lower extremity strength, and functional capacity through walking and sit to stand test.
Change in physical performance assessed by hand grip strength. | 52 weeks
  Grip strength is measured on the dominant hand with a hydraulic hand-held dynamometer.
Change in cognitive function assessed using the Repeatable Battery for the Assessment of Neuropsychological Status (RBANS) test battery. | 52 weeks
  The RBANS test battery is composed of tests on immediate memory, visuospatial/constructional abilities, language, attention, and delayed memory. Score range: 40-160. A higher score indicates a better performance.

OTHER OUTCOMES:
Change in daily step count. | 52 weeks
  Measured in number of steps using Axivity wearable sensors. Counts the total number of steps taken by an individual over a specified period.
Change in overall activity level. | 52 weeks
  Measured in activity counts using Axivity's accelerometer data. Quantifies the total amount of physical activity based on intensity and duration.
Change in speed of movements. | 52 weeks
  Measured in per second (m/s) using Axivity's accelerometer and gyroscope data. Calculates the average or peak speed of movements during different activities.
Change in acceleration of movements. | 52 weeks
  Measured in meters per second squared (m/s2) using Axivity's accelerometer data. Measures the rate of change of speed, indicating how quickly an individual is increasing or decreasing speed during activities. Measured in meters per second squared (m/s^2) using Axivity's accelerometer data.
Change in angular velocity of movements. | 52 weeks
  Measured in radians per second (rad/s) using Axivity's gyroscope data. Measures the rate of rotation around an axis, assessing movement dynamics.
Change in Activities of Daily Living (ADL) score. | 52 weeks
  Assessed by the Barthel Index Activities of Daily Living (ADL) scale. Score range: 0 - 20. A higher score indicate better functional status.
Change in Independent living skills (IADL) score. | 52 weeks
  Assessed by the Nottingham Instrumental Activities of Daily Living (IADL) scale. Score range: 0-66. A higher score indicate better functional status.
Change in mobility assessed by the Life Space Questionnaire (LSQ). | 52 weeks
  Score range: 0-18. A higher score indicates more limited mobility.
Change in mood assessed by the Montgomery Aasberg Depression Rating Scale (MADRS). | 52 weeks
  Score range: 0-54. Higher score indicates a greater severity of depressive symptoms.
Change in self-reported mood assessed by the Geriatric depression scale (GDS). | 52 weeks
  Score range: 0-30. A higher score indicates more severe depressive symptoms.
Change in self-assessment of perceived health assessed by the Short form 36 (RAND-36). | 52 weeks
  The RAND-36 assessment does not provide a single summary score; rather, it offers scores for each of eight domains (physical functioning, role limitations due to physical health problems, role limitations due to personal or emotional problems, emotional well-being, social functioning, energy/fatigue, pain, and general health perceptions), allowing for a comprehensive assessment of a person's health-related quality of life.
Change in sleep assessed by the Pittsburgh Sleep Quality Index (PSQI) global score. | 52 weeks
  Seven component scores are derived, each scored 0 (no difficulty) to 3 (severe difficulty). The component scores are summed to produce a global score (range 0 to 21). Higher scores indicates worse sleep quality.
Change in smell identification capacity assessed using the Brief Smell Identification Test (BSIT). | 52 weeks
  Score range: 0-12. A higher score indicates better smell identification.
Change in nutritional status assessed using the Mini Nutritional Assessment (MNA) form. | 52 weeks
  Score range: 0-30. A higher score indicates better nutritional status.
Change in sarcopenia assessment. | 52 weeks
  Assessed using anthropometric measures (weight and height will be combined to report BMI in kg/m^2).
Change in health-related quality of life assessed by a standardized measure of quality of life (the EQ-5D-5L questionnaire). | 52 weeks
  The EQ-5D-5L does not provide a single summary score; rather, it offers three levels, where level 1 indicates higher quality of life.
Change in cognitive function using the Grooved Pegboard test. | 52 weeks
  Test on motor function, attention, and executive functioning.
Change in cumulative illness / comorbidity examined using the Cumulative Illness Rating Scale-Geriatric (CIRS-G). | 52 weeks
  CIRS-G does not provide a single summary score; rather, it offers four levels of severity where level 4 is the highest severity of comorbidity.
Change in social support assessed using the Multidimensional scale of perceived social support (MSPSS). | 52 weeks
  Score range: 12-84. Higher scores indicates higher perceived support.
The between-visit difference in cerebral NAD levels. | 52 weeks
  Measured by 31P-Magnetic resonance spectroscopy (31P-MRS)
The between-visit difference in expression of the Nicotinamide Riboside Related Pattern (NRRP). | 52 weeks
  Measured by fluorodeoxyglucose (FDG)-positron emission tomography (FDG-PET).
The between-visit difference in levels of NAD-metabolites in whole blood. | 52 weeks
  Measured by liquid chromatography-mass spectrometry (LC-MS).
Change in blood-based biomarkers. | 52 weeks
  Blood routine biochemistry encompassing cardiovascular-, metabolic-, renal- and hepatic markers, immune- and inflammatory profiles.
Change in gene and protein expression levels related to lysosomal and proteasomal function. | 52 weeks
  The between-visit change in gene and protein expression levels related to lysosomal and proteasomal function in whole blood, measured by RNA sequencing (RNAseq) and proteomics (LC-MS), respectively.
Change in genomic distribution of DNA methylation. | 52 weeks
  The between-visit difference in genomic distribution of DNA methylation, measured by the Illumina Infinium MethylationEPIC Kit.
Change in levels of DNA methylation. | 52 weeks
  The between-visit difference in levels of DNA methylation, measured by the Illumina Infinium MethylationEPIC Kit.
Change in gut microbiome composition. | 52 weeks
  The between-visit difference in gut microbiome composition, assessed by metagenomics in fecal samples.
Change in fecal metabolomics. | 52 weeks
  The between-visit difference in fecal metabolomics, including fatty acid profiling.
Change in levels of inflammatory cytokines in serum. | 52 weeks
  The between-visit difference in levels of inflammatory cytokines in serum measured using the ELISA method.

CONTACTS AND LOCATIONS:
Overall Officials: Charalampos Tzoulis, PhD, Study Director — Haukeland University Hospital
Locations (2):
- Norway (2):
  - Haukeland University Hospital, Bergen, Vestland
  - Haukeland University Hospital, Bergen

IPD SHARING:
Plan to Share IPD: No